CLINICAL TRIAL: NCT00102076
Title: Implementing the Assent Requirement for Research With Children
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020054; 02-CC-0054
Record Dates: First submitted 2005-01-19; First posted 2005-01-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-09-18

CONDITIONS: Healthy
Keywords: Minimal; Risk; Regulations; Parents; IRB; Surgery; Assent Requirement

SUMMARY:
One of the principal safeguards mandated by the Federal Regulations governing clinical research with children is the assent requirement: children who are capable must provide an affirmative agreement to participate unless the research "holds out a prospect of direct benefit that is important to the health or well-being of the children and is available only in the context of the research" (46.408). Despite the importance of the assent requirement, the Federal regulations offer no guidelines on its implementation. In the present study, we propose to survey children and one of their parents in order to obtain information concerning children's role in making decisions concerning their participation in clinical research. Five elements of children's involvement in the decision-making process with respect to their participation in clinical research will be assessed: 1) receipt of information concerning the available options; 2) understanding of this information; 3) assessment of the available options; 4) expression of a preferred option; and 5) coordination with parental decision-making.

Three groups will be enrolled: 1. Minor/Parent pairs where the minor is participating in, or is in follow-up for, a drug treatment research study for cancer 2. Minor/Parent pairs where the minor is participating in, or is in follow-up for, a drug treatment research study for asthma, and 3. Minor/Parent pairs where the minor is receiving on-going clinical care for asthma. Children 7-14 years of age will be enrolled. Total enrollment will be 400 subject pairs, approximately 150 in cancer research, 150 in asthma research and 100 involved in clinical care for asthma, with approximate balance between the sites. Two formalized survey instruments - research/clinical minor, research/clinical parent - will be developed in consultation with Research Triangle Institute (RTI).

DETAILED DESCRIPTION:
One of the principal safeguards mandated by the Federal Regulations governing clinical research with children is the assent requirement: children who are capable must provide an affirmative agreement to participate unless the research "holds out a prospect of direct benefit that is important to the health or well-being of the children and is available only in the context of the research" (46.408). Despite the importance of the assent requirement, the Federal regulations offer no guidelines on its implementation. In the present study, we propose to survey children and one of their parents in order to obtain information concerning children's role in making decisions concerning their participation in clinical research. Five elements of children's involvement in the decision-making process with respect to their participation in clinical research will be assessed: 1) receipt of information concerning the available options; 2) understanding of this information; 3) assessment of the available options; 4) expression of a preferred option; and 5) coordination with parental decision-making.

Three groups will be enrolled: 1. Minor/Parent pairs where the minor is participating in, or is in follow-up for, a drug treatment research study for cancer 2. Minor/Parent pairs where the minor is participating in, or is in follow-up for, a drug treatment research study for asthma, and 3. Minor/Parent pairs where the minor is receiving on-going clinical care for asthma. Children 7-14 years of age will be enrolled. Total enrollment will be 400 subject pairs, approximately 150 in cancer research, 150 in asthma research and 100 involved in clinical care for asthma, with approximate balance between the sites. Two formalized survey instruments - research/clinical minor, research/clinical parent - will be developed in consultation with Research Triangle Institute (RTI).

ELIGIBILITY:
* INCLUSION CRITERIA:

Children in Research Studies:

* Currently enrolled in an ongoing medical intervention protocol, including follow-up, for cancer or asthma at one of the participating sites.
* Post initial visit.
* Enrolled within the previous year.
* Physically and cognitively able to participate in a 30 minute interview.
* Ability to understand and speak English.
* Age 7-14.

Parents of Children in Research Studies:

* Parent of an eligible research child.
* Physically and cognitively able to participate in a 30 minute interview.
* Ability to understand and speak English.

Children Receiving Clinical Care:

* Receiving clinical care at a clinic at one of the participating sites for cancer or asthma.
* Post initial visit.
* Physically and cognitively able to participate in a 30 minute interview.
* Ability to understand and speak English.
* Age 7-14.

Parents of Children Receiving Care:

* Parent of an eligible clinical minor.
* Physically and cognitively able to participate in a 30 minute interview.
* Ability to understand and speak English.

EXCLUSION CRITERIA:

Inability to speak English.

Inability to understand spoken English.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800
Dates: Start 2001-11-16; Study Completion 2006-09-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States